CLINICAL TRIAL: NCT07320027
Title: Comparison of the Acute Effects of Static Stretching, Dynamic Stretching, and Proprioceptive Exercises on Proprioception, Muscle Strength, Balance, and Explosive Power: A Randomized Controlled Trial.
Brief Title: Acute Impact of Static, Dynamic, and Proprioceptive Exercises on Proprioception, Strength, Balance, and Explosive Power
Acronym: SSDSPE-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Muhammet Talha DOĞAN, Principal Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22817
Record Dates: First submitted 2025-08-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Control; Balance; Musculoskeletal Function
Keywords: Proprioception; Static stretching; Dynamic stretching; Balance; Explosive Power

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioception group (Experimental): The group that received proprioception exercises
  Interventions: Other: Proprioceptive Exercise Group
- Dynamic tension group (Experimental): The group that received dynamic stretching exercises
  Interventions: Other: Dynamic Stretching Exercise Group
- Static tension group (Experimental): The group that received static stretching exercises
  Interventions: Other: Static Stretching Exercise Group

INTERVENTIONS:
Other: Static Stretching Exercise Group — Our exercise group where we applied the static stretching protocol
  Other Names: SG
  Arms: Static tension group
Other: Dynamic Stretching Exercise Group — Our exercise group where we applied the dynamic stretching protocol
  Other Names: DG
  Arms: Dynamic tension group
Other: Proprioceptive Exercise Group — Proprioceptive Exercise Program
  Other Names: PG
  Arms: Proprioception group

SUMMARY:
The purpose of this randomized controlled trial is to compare the acute effects of static stretching, dynamic stretching, and proprioceptive exercises on proprioception, muscle strength, balance, and explosive power in young athletes. The study aims to determine how different stretching and exercise modalities influence short-term performance parameters.

The primary questions this study aims to answer are:

Do static stretching, dynamic stretching, and proprioceptive exercises have different acute effects on proprioception?

Do these interventions cause different changes in muscle strength, balance, and explosive power?

Researchers will compare the static stretching, dynamic stretching, and proprioceptive exercise groups to determine which method produces greater improvements in the measured performance parameters.

Participants will:

Perform one of the three assigned exercise protocols according to a standardized warm-up procedure

Undergo pre- and post-exercise assessments, including:

Proprioception (measured with an isokinetic device)

Muscle strength (measured with an isokinetic device)

Balance (measured with a Y balance test and BESS balance test)

Explosive power (measured with the Sargent Vertical Jump Test)

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the acute effects of static stretching, dynamic stretching, and proprioceptive exercises on knee joint position sense (proprioception), muscle strength, balance, and explosive power in young male soccer players.

Proprioception, the ability to sense the position and movement of joints, muscles, and tendons, plays a critical role in maintaining joint stability. Proprioceptive exercises are widely used among athletes to enhance performance and reduce injury risk. Stretching exercises, particularly static and dynamic techniques, are commonly integrated into warm-up routines to improve flexibility, joint range of motion, and neuromuscular function. However, direct comparisons of the acute effects of static stretching, dynamic stretching, and proprioceptive exercises remain limited.

In this study, healthy male soccer players aged 14-19 years, with at least five years of competitive experience, no knee pain in the past two months, and no history of knee surgery, will be included. Participants will be randomly assigned (block randomization) into three groups:

Static Stretching Group - A controlled-position protocol targeting the quadriceps, hamstrings, plantar flexors, and dorsiflexors, with specific hold durations.

Dynamic Stretching Group - A repetitive movement protocol for the same muscle groups, with gradual speed increases.

Proprioceptive Exercise Group - A 10-exercise proprioceptive training program performed on a BOSU ball, focusing on lower-limb awareness, postural control, and dynamic balance.

All groups will perform a standardized 10-minute warm-up on a cycle ergometer before their respective protocols.

Assessments will be conducted before and immediately after the intervention:

Knee joint position sense (proprioception) - measured with an ISOMED 2000 isokinetic dynamometer

Muscle strength - isokinetic testing of knee flexors and extensors using the isokinetic device

Static balance - Balance Error Scoring System (BESS) test

Dynamic balance - Y-Balance Test

Explosive power - Sargent Vertical Jump Test

The primary hypothesis is that proprioceptive exercises will produce greater acute improvements in proprioception, balance, and explosive power, while dynamic stretching may yield higher acute gains in muscle strength. Findings from this study are expected to inform evidence-based warm-up and training strategies for young soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Playing football for at least 5 years.
* Not experiencing knee pain for the last 2 months.
* No history of knee surgery.
* Practicing for 90 minutes at least 5 days a week.
* Volunteering to participate in the study.
* Being between 14 and 19 years old.

Exclusion Criteria:

* Having experienced knee pain for the last two months.
* Having had knee surgery.
* Not willing to participate.

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 48 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Knee Joint Position Sense Error (degrees) | Baseline and 1 day
  Angular joint position matching error (degrees) measured using the ISOMED 2000 isokinetic dynamometer with passive reproduction of target angles.
Peak Torque during Knee Extension (Nm) | Baseline and 1 day
  Peak torque (Nm) during knee extension assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.

SECONDARY OUTCOMES:
Peak Torque during Knee Flexion (Nm) | Baseline and 1 day
  Peak torque (Nm) during knee flexion assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Total Work during Knee Extension (J) | Baseline and 1 day
  Total work (J) produced during knee extension assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Total Work during Knee Flexion (J) | Baseline and 1 day
  Total work (J) produced during knee flexion assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Average Work during Knee Extension (J) | Baseline and 1 day
  Average work (J) during knee extension assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Average Work during Knee Flexion (J) | Baseline and 1 day
  Average work (J) during knee flexion assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Maximum Work during Knee Extension (J) | Baseline and 1 day
  Maximum work (J) during knee extension assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Maximum Work during Knee Flexion (J) | Baseline and 1 day
  Maximum work (J) during knee flexion assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Average Power during Knee Extension (W) | Baseline and 1 day
  Average power (W) during knee extension assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Average Power during Knee Flexion (W) | Baseline and 1 day
  verage power (W) during knee flexion assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Knee Joint Angle at Peak Torque during Extension (degrees) | Baseline and 1 day
  The knee joint angle (degrees) at which peak torque occurs during knee extension, assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Knee Joint Angle at Peak Torque during Flexion (degrees) | Baseline and 1 day
  The knee joint angle (degrees) at which peak torque occurs during knee flexion, assessed using the ISOMED 2000 isokinetic dynamometer. Testing was performed in concentric mode at 60 deg/s.
Y Balance Test Composite Score (percent) | Baseline and 1 day
  Dynamic balance performance evaluated using the normalized composite reach score from the Y Balance Test (percent).
BESS Total Error Score (points) | Baseline and 1 day
  Static balance performance measured using the Balance Error Scoring System (BESS); higher scores indicate worse balance.
Vertical Jump Height (cm) - Sargent Test | Baseline and 1 day
  Explosive lower-limb power measured using the Sargent Vertical Jump Test (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan ALTUNTAŞ YILMAZ E Dr. Öğr. Üyesi, Doctor, Study Director — Necmettin Erbakan University
Locations (1):
- Tümosan Konyaspor Facilities, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stehouwer CD. [Hormonal supplements for postmenopausal women: no evidence of protection against cardiovascular disease]. Ned Tijdschr Geneeskd. 2001 Jan 13;145(2):61-4. Dutch. PMID 11225257